CLINICAL TRIAL: NCT06688214
Title: Effects of Kinesio Taping and Scapular Stabilization Exercises on ROM, Pain and Function in Badminton Players With Subacromial Impingement Syndrome
Brief Title: Effects of KT and Scapular Stabilization Exercises.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0424
Record Dates: First submitted 2024-10-27; First posted 2024-11-14 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Subacromial Impingement; Kinesiotaping; scapular exercises; shoulder rehabilitation; Rotator cuff muscles
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kinesio Taping (Experimental): Kinesio Taping treatment
  Interventions: Other: Kinesio Taping treatment
- Scapular Stabilization Exercises (Active Comparator): Scapular Stabilization Exercises
  Interventions: Other: Scapular Stabilization Exercises

INTERVENTIONS:
Other: Kinesio Taping treatment — Therapeutic KT application administered to patients in group A. The KT treatment was completed in compliance with Kase's recommended methodology for rotator cuff tendinitis/impingement. Initially, an inhibitory approach was used to apply a supraspinatus Y-strip from its insertion to its origin. The measurement of the strip's length was taken from the acromion to the scapular spine. The base of the strip was later applied to the tuberculum major while the patient was seated; the superior tale of the Y-strip was then terminated at the superomedial angle of the scapula, passing between the middle and superior fibers of the trapezius with light tension (% 15-25); the shoulder was then extended, adducted, and internally rotated with cervical contralateral bending; the final portion of the tape (2.5-5 cm) was applied painlessly.
  Arms: Kinesio Taping
Other: Scapular Stabilization Exercises — Participants in Group B engage in a twice-weekly, supervised SSE exercise program that is based on the clinical decision algorithm that has been recommended by an expert panel. The goal of scapular orientation training was to normalize the scapula's resting posture and enhance proprioception. Subsequently, three scapular control exercises were executed: a closed kinetic chain exercise known as the "unilateral bench press," bilateral shoulder flexion up to 60°, and a scapular control exercise including bilateral shoulder retraction and extension in the prone position. There was no discomfort involved in performing the exercises, and each session may consist of no more than four exercises. The dosage and progressions were based on the objectives of each exercise; each exercise was performed 8-10 times with a 5- to 10-second hold in between, and there was a 30-to 1-minute rest period.
  Arms: Scapular Stabilization Exercises

SUMMARY:
The distance between the acromion bone and the head of the humerus narrows in subacromial impingement syndrome. This narrowing leads to the compression of sensitive structures and results in pain and decreased functional performance.While taping and scapular stabilizing exercises are commonly used in the treatment of subacromial impingement syndrome, no comparisons were conducted previously between their effectiveness.

This randomized clinical trial will be conducted at Punjab Sports Board, Lahore.This study will include patients with age group ≥18 years; pain located on the anterolateral side of the shoulder for ≥3 months with positive clinical signs.

Group A will receive Kinesiotaping protocol and Group B will receive Scapular Stabilization exercises protocol.

DETAILED DESCRIPTION:
The distance between the acromion bone and the head of the humerus narrows in subacromial impingement syndrome. This narrowing leads to the compression of sensitive structures and results in pain and decreased functional performance. Subacromial Impingement syndrome can be Primary and Secondary, both types could present patterns of postural deviation, painful arc, and altered biomechanics of muscles.While taping and scapular stabilizing exercises are commonly used in the treatment of subacromial impingement syndrome, no comparisons were conducted previously between their effectiveness.

This randomized clinical trial will be conducted at Punjab Sports Board, Lahore. This study will include patients with age group ≥18 years; pain located on the anterolateral side of the shoulder for ≥3 months with positive clinical signs of SIS, such as the Neer or Hawkins-Kennedy test, a painful arc, pain on resisted external rotation, or the Empty Can test after exclusion of cervical radiculopathy, osteoarthritis in the acromioclavicular or glenohumeral joint, calcific tendinitis, adhesive capsulitis, glenohumeral instability or a partial or full-thickness rotator cuff tear, clinical history of acute trauma, previous surgery or previous fracture in the affected shoulder; or corticosteroid injection into the shoulder joint in the previous 12 months.Participants will be divided into two groups. Group A will receive Kinesio-taping protocol and Group B will receive Scapular Stabilization exercises protocol.Patients will be assessed Shoulder Pain And Disability Index (SPADI). Changes in upper limb function Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire. Pain intensity {Visual Analog Scale (VAS) Kinesiophobia {Tampa Scale of Kinesiophobia (TSK)}. The findings can contribute to the growing evidence based supporting whether the use of Kinesio taping or scapular stabilization Exercises improve ROM, 5 Pain and function in patients with Subacromial impingement syndrome. Analysis will be done by statistical package for social sciences SPSS 29.

ELIGIBILITY:
Inclusion Criteria:

Participants with age between 18 to 55 years. Participants with pain on the anterolateral side of the shoulder for ≥3 months. Participants diagnosed with ≥3 positive clinical signs of SIS, such as the Neer or Hawkins-Kennedy test, a painful arc by a sports physical therapist.

Mild or Moderate pain on resisted external rotation, or the Empty Can test.

Exclusion Criteria:

Diagnosis of cervical radiculopathy. Participants with osteoarthritis in the acromioclavicular or glenohumeral joint.

Calcific tendinitis, adhesive capsulitis, glenohumeral instability or a partial or full-thickness rotator cuff tear, clinical history of acute trauma, previous surgery or previous fracture in the affected shoulder. Corticosteroid injection into the shoulder joint in the previous 12 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain And Disability Index (SPADI). | 1 week
  In order to assess the level of pain and impairment, established the shoulder pain and disability index, which modified. It has thirteen questions total, split into two auxiliary scales: five questions measure pain intensity, and eight questions assess upper limb disability when completing various activities of daily living. The pain subscale has five questions. A 10-point Likert scale was used to rate the thirteen things, with 0 denoting no discomfort and 10 denoting extremely severe pain. Each tool's results were transformed into a 100-point rating system. The degree of shoulder pain, injury, and disability increases with the tool's score.
Changes in upper limb function Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | 1 week
  The Spanish version of the Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire was used to measure upper limb function. Scores range from 0 to 100 points, with higher scores indicating poorer function.The MCID is 11 points.Patients were asked to fill out DASH questionnaires, to apply marks to the point that they felt represented their perception of their current state
Pain intensity {Visual Analog Scale (NPRS). | 1 week
  The numeric pain rating scale for pain (NPRS) is generally captured on a 10- centimeter line, with 0 representing no pain, 5 indicating moderate pain, and 10 representing worst possible pain. Michener and colleagues15 reported that the minimally clinically important difference (MCID) for the NPRS was 2.17 for subjects with shoulder pain due to both surgical and non-surgical sources
Kinesiophobia {Tampa Scale of Kinesiophobia (TSK) | 1 week
  The original 17-item Tampa Scale of Kinesiophobia (TSK) was used to assess pain- related fear of movement. The scores range from 17 to 68 points, with higher scores indicating greater fear of movement and or (re-)injury. The MCID for people with chronic pain is 5.6 points; however, the MCID for people with SIS or rotator cuff disease has not been established.
Standard Goniometer | 1 week
  Shoulder flexibility was measured using a standard goniometer, which has a reported accuracy within 1° and a range of 180°. Goniometry is a common clinical method used for measuring shoulder complex ROM associated with adequate reliability.A standard goniometer is used to evaluate the passive range of motion of all joints of the shoulder girdle and upper limb. Deficits of joint motion from immobility result in contracture of the joint capsule, adhesions in the joints, and shortening of both muscle and tendons above the affected joints

CONTACTS AND LOCATIONS:
Overall Officials: Imran Ghafoor Dr., DPT,M.phil, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goksu H, Tuncay F, Borman P. The comparative efficacy of kinesio taping and local injection therapy in patients with subacromial impingement syndrome. Acta Orthop Traumatol Turc. 2016 Oct;50(5):483-488. doi: 10.1016/j.aott.2016.08.015. Epub 2016 Sep 23. PMID 27670388
- [Background] Kul A, Ugur M. Comparison of the Efficacy of Conventional Physical Therapy Modalities and Kinesio Taping Treatments in Shoulder Impingement Syndrome. Eurasian J Med. 2019 Jun;51(2):139-144. doi: 10.5152/eurasianjmed.2018.17421. Epub 2018 Nov 30. PMID 31258353
- [Background] Ravichandran H, Janakiraman B, Gelaw AY, Fisseha B, Sundaram S, Sharma HR. Effect of scapular stabilization exercise program in patients with subacromial impingement syndrome: a systematic review. J Exerc Rehabil. 2020 Jun 30;16(3):216-226. doi: 10.12965/jer.2040256.128. eCollection 2020 Jun. PMID 32724778
- [Background] Sharma S, Ghrouz AK, Hussain ME, Sharma S, Aldabbas M, Ansari S. Progressive Resistance Exercises plus Manual Therapy Is Effective in Improving Isometric Strength in Overhead Athletes with Shoulder Impingement Syndrome: A Randomized Controlled Trial. Biomed Res Int. 2021 Jun 30;2021:9945775. doi: 10.1155/2021/9945775. eCollection 2021. PMID 34307681
- See also: Progressive Resistance Exercises plus Manual Therapy Is Effective in Improving Isometric Strength in Overhead Athletes with Shoulder Impingement Syndrome: A Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/34307681
- See also: Effect of scapular stabilization exercise program in patients with subacromial impingement syndrome: a systematic review — https://pubmed.ncbi.nlm.nih.gov/32724778
- See also: Effectiveness of Scapular Stabilization Versus Non-Stabilization Stretching on Shoulder Range of Motion, a Randomized Clinical Trial — https://pubmed.ncbi.nlm.nih.gov/35693853
- See also: Comparison of the Efficacy of Conventional Physical Therapy Modalities and Kinesio Taping Treatments in Shoulder Impingement Syndrome — https://pubmed.ncbi.nlm.nih.gov/31258353
- See also: The comparative efficacy of kinesio taping and local injection therapy in patients with subacromial impingement syndrome — https://pubmed.ncbi.nlm.nih.gov/27670388